CLINICAL TRIAL: NCT04968626
Title: Relationship Between Spinopelvic Parameters and Clinical Symptoms of Low-grade Lumbar Isthmic Spondylolisthesis: a Retrospective Analysis
Brief Title: Relationship Between Spinopelvic Parameters and Clinical Symptoms of Low-grade Lumbar Isthmic Spondylolisthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M2019125
Record Dates: First submitted 2021-06-27; First posted 2021-07-20 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2020-03

CONDITIONS: Isthmic Spondylolisthesis
Keywords: Isthmic Spondylolisthesis; Spinopelvic parameter; Clinical symptom; Pelvic incidence; Lumbar lordosis
MeSH Terms: conditions — Lordosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IS GROUP (Experimental): Patients who received an operation to treat their isthmic spondylolisthesis (IS, Meyerding grade I-II)
  Interventions: Radiation: PI-LL
- AS GROUP (No Intervention): The asymptomatic adults had no history of severe back pain or spinal trauma

INTERVENTIONS:
Radiation: PI-LL — The pelvic parameters were collected including PI, pelvic tilt (PT), sacral slope (SS) and LL ,and compared between IS patients and the AS group. Besides, spinopelvic malalignment was defined as an absolute value of PI-LL greater than 10.In the IS group,the clinical symptoms were assessed with the Japanese Orthopaedic Association (JOA) score and the visual analogue scale (VAS). We compared spinopelvic parameters between the asymptomatic adults and the IS patients. Additionally, we investigated correlations between spinopelvic parameters and clinical symptoms.
  Other Names: PI-LL mismatch
  Arms: IS GROUP

SUMMARY:
This was a retrospective study.PI and LL greatly influence IS and its progression. However, relationships between the spinopelvic parameters and clinical symptoms of patients with IS were not fully investigated in previous studies. Investigators hypothesized that spinopelvic parameters might be related to the clinical symptoms of IS patients. Therefore, the purpose of the present study was to investigate whether differences in spinopelvic parameters, especially spinopelvic alignment, may be associated with the clinical symptoms of low-grade IS patients.

DETAILED DESCRIPTION:
Isthmic spondylolisthesis (IS) is one of the most common types of spondylolisthesis, and spinopelvic parameters are closely related to the clinical symptoms of spinal diseases. In this study, investigators attempted to investigate the relationship between spinopelvic parameters and clinical symptoms of patients with low-grade (Meyerding grade I-II) isthmic spondylolisthesis (IS).

A total of 120 patients with low-grade IS and 106 asymptomatic adults were included in this study. Sex, age and body mass index (BMI) were also collected. Various spinopelvic parameters were evaluated in whole-spine standing-position X-rays. The following spinopelvic parameters were measured: pelvic incidence (PI), sacral slope (SS), pelvic tilt (PT) and lumbar lordosis (LL). The clinical symptoms of the IS patients were assessed with the Japanese Orthopaedic Association (JOA) score and the visual analogue scale (VAS). Investigators compared spinopelvic parameters between the asymptomatic adults and the IS patients. Additionally, investigators investigated correlations between spinopelvic parameters and clinical symptoms.

ELIGIBILITY:
Inclusion Criteria:

* isthmic spondylolisthesis subjects had spondylolisthesis at L4 or L5 (Meyerding grade I-II) with whole-spine standing lateral images

Exclusion Criteria:

* spondylolisthesis of other types (Degenerative, dysplastic, etc.);
* Lumbar infection and/or tumor diseases;
* A previous history of lumbar fusion surgery.

Ages: 54 Years to 76 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2019-03-19 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
PI | through study completion, an average of 1 year
  pelvic incidence
SS | through study completion, an average of 1 year
  sacral slope
PT | through study completion, an average of 1 year
  pelvic tilt
LL | through study completion, an average of 1 year
  lumbar lordosis
PI-LL | through study completion, an average of 1 year
  pelvic incidence minus lumbar lordosis

SECONDARY OUTCOMES:
VAS | through study completion, an average of 1 year
  visual analogue scale
JOA | through study completion, an average of 1 year
  The Japanese Orthopaedic Association (JOA)

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Result] Randall RM, Silverstein M, Goodwin R. Review of Pediatric Spondylolysis and Spondylolisthesis. Sports Med Arthrosc Rev. 2016 Dec;24(4):184-187. doi: 10.1097/JSA.0000000000000127. PMID 27811518
- [Result] Urrutia J, Cuellar J, Zamora T. Spondylolysis and spina bifida occulta in pediatric patients: prevalence study using computed tomography as a screening method. Eur Spine J. 2016 Feb;25(2):590-5. doi: 10.1007/s00586-014-3480-y. Epub 2014 Jul 29. PMID 25070790
- [Result] Ramadorai U, Hire J, DeVine JG, Brodt ED, Dettori JR. Incidental findings on magnetic resonance imaging of the spine in the asymptomatic pediatric population: a systematic review. Evid Based Spine Care J. 2014 Oct;5(2):95-100. doi: 10.1055/s-0034-1386753. PMID 25278883
- [Result] Beutler WJ, Fredrickson BE, Murtland A, Sweeney CA, Grant WD, Baker D. The natural history of spondylolysis and spondylolisthesis: 45-year follow-up evaluation. Spine (Phila Pa 1976). 2003 May 15;28(10):1027-35; discussion 1035. doi: 10.1097/01.BRS.0000061992.98108.A0. PMID 12768144
- [Result] Duval-Beaupere G, Schmidt C, Cosson P. A Barycentremetric study of the sagittal shape of spine and pelvis: the conditions required for an economic standing position. Ann Biomed Eng. 1992;20(4):451-62. doi: 10.1007/BF02368136. PMID 1510296
- [Result] Maciejczak A, Jablonska K, Baczek D, Barnas P, Czternastek M, Dudziak P, Georgiew F, Jagiello-Bajer B, Litwora B, Maslanka P, Konior R, Orzech J. Changes in spino-pelvic alignment after surgical treatment of isthmic spondylolisthesis. Neurol Neurochir Pol. 2014 Jan-Feb;48(1):21-9. doi: 10.1016/j.pjnns.2013.05.001. Epub 2014 Jan 23. PMID 24636766
- [Result] Park SJ, Lee CS, Chung SS, Kang KC, Shin SK. Postoperative changes in pelvic parameters and sagittal balance in adult isthmic spondylolisthesis. Neurosurgery. 2011 Jun;68(2 Suppl Operative):355-63; discussion 362-3. doi: 10.1227/NEU.0b013e3182117249. PMID 21336205
- [Result] Lafage R, Liabaud B, Diebo BG, Oren JH, Vira S, Pesenti S, Protopsaltis TS, Errico TJ, Schwab FJ, Lafage V. Defining the Role of the Lower Limbs in Compensating for Sagittal Malalignment. Spine (Phila Pa 1976). 2017 Nov 15;42(22):E1282-E1288. doi: 10.1097/BRS.0000000000002157. PMID 28306639
- [Result] Minamide A, Yoshida M, Iwahashi H, Simpson AK, Yamada H, Hashizume H, Nakagawa Y, Iwasaki H, Tsutsui S, Kagotani R, Sonekatsu M, Sasaki T, Shinto K, Deguchi T. Minimally invasive decompression surgery for lumbar spinal stenosis with degenerative scoliosis: Predictive factors of radiographic and clinical outcomes. J Orthop Sci. 2017 May;22(3):377-383. doi: 10.1016/j.jos.2016.12.022. Epub 2017 Feb 1. PMID 28161236
- [Result] Shi L, Chen Y, Miao J, Shi J, Chen D. Reduction of Slippage Influences Surgical Outcomes of Grade II and III Lumbar Isthmic Spondylolisthesis. World Neurosurg. 2018 Dec;120:e1017-e1023. doi: 10.1016/j.wneu.2018.08.217. Epub 2018 Sep 7. PMID 30201580